CLINICAL TRIAL: NCT04955132
Title: Impact of E-learning on Parental Confidence in Managing Food Allergy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Vilnius University (Other)
Responsible Party: Principal Investigator, Ieva Adomaite, Principal Investigator, Vilnius University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 18BMTV33
Record Dates: First submitted 2021-07-03; First posted 2021-07-08 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Food Allergy in Children; Food Allergy in Infants
Keywords: Food allergy; Milk; Egg; Wheat; Children
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-learning (Experimental): Participants (parents of food-allergic children) will use an E-learning platform on food allergies for one month.
  Interventions: Behavioral: E-learning
- Standard care (No Intervention): Participants (parents of food-allergic children) will receive standard allergist consulting.

INTERVENTIONS:
Behavioral: E-learning — The participants in the experimental arm will be able to use a food allergy e-learning tool, that provides comprehensive knowledge of the most common food allergies (milk, egg and wheat), their management and dietary guidelines.
  Arms: E-learning

SUMMARY:
Education and dietary support are integral in managing food allergy in children. The study aim is to analyze the impact of E-learning on parental confidence in managing their child's food allergy.

DETAILED DESCRIPTION:
Food allergy is a common childhood morbidity, that has increased in prevalence over the last few decades. Education and dietary support is integral in managing food allergy in children; however it is labor intensive and requires financial resources, which places an economic burden on the healthcare system. The study aim is analyze the impact of E-learning on parental confidence in managing their child's food allergy.

ELIGIBILITY:
Inclusion Criteria:

* Legal caregivers of a child that is allergic (confirmed by an allergist) to at least one of the main food allergens (cow's milk, egg or wheat) and is following an elimination diet to at least one of these allergens.
* Internet access available.

Exclusion Criteria:

* Participant non proficient in Lithuanian.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Parental confidence in managing food allergy | After 1 month.
  Parental confidence will be assessed using Food Allergy Self-Efficacy Scale for Parents (FASE-P). Single item minimum score - 0, maximum score - 100. Higher scores represent higher parental confidence.

SECONDARY OUTCOMES:
Parental satisfaction | After 1 month.
  Parental satisfaction will be assessed using Visual Analog Satisfaction Scale. Minimum score - 0, maximum score - 100. Higher score represents higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ieva Adomaite, Principal Investigator — Vilnius University Faculty of Medicine
Locations (1):
- Vilnius University Hospital Santaros Clinics, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Yes
All collected data, following deidentification will be available.
Supporting Information: Study Protocol, SAP, Analytic Code